CLINICAL TRIAL: NCT01087671
Title: Ocular Signs and Symptoms in Patients With Ocular Hypertension or Open-angle Glaucoma Switched From Preserved Latanoprost 0.005% Eye Drops to Preservative Free Tafluprost Eye Drops
Brief Title: Ocular Signs and Symptoms in Glaucoma Patients Switched From Latanoprost to Preservative Free Tafluprost Eye Drops
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 77553
Record Dates: First submitted 2010-03-03; First posted 2010-03-16 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2010-11

CONDITIONS: Ocular Hypertension; Open-Angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — tafluprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-lable study with one arm (Other)
  Interventions: Drug: tafluprost

INTERVENTIONS:
Drug: tafluprost — prostaglandin analogue

SUMMARY:
The purpose of this study is to investigate if changes in ocular signs and symptoms occur in patients with ocular hypertension or glaucoma when they switch from latanoprost 0.005% (Xalatan) to preservative free Tafluprost eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of ocular hypertension or open angle glaucoma for which the patient has been using latanoprost 0.005% as his/her prior medication.
* Evaluable patients must have ocular surface related symptoms and/or signs with their prior medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in ocular symptoms and signs | From Screening (Visit 1) to12 weeks.
  Ocular symptoms include: irritation/burning/stinging, foreign body sensation, tearing, itching and dry eye sensation.
  Following signs will be evaluated: tear break-up time, corneal and conjunctival fluorescein staining, blepharitis, conjunctival redness and tear secretion (schirmer test).

SECONDARY OUTCOMES:
Secondary outcome measures include the assessment of safety and quality of life parameters. | From Screening (visit 1) to 12 weeks
  Safety parameters include: best-corrected visual acuity, biomicroscopy, ophthalmoscopy, visual field test, drop discomfort upon instillation, intra ocular pressure, quality of life and adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Evgeniy Egorov, Professor, Principal Investigator — State Educational Establishment of Higher Professional Education "Russian State Medical University of Federal Service on Surveillance in Healthcare and Social Development of Russian Federation"